CLINICAL TRIAL: NCT04118569
Title: Personalized Experiences to Inform Improved Communication for Patients With Life Limiting Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-1874; 4R00NR016686-03 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure; Renal Failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: 50% of patient participants will complete the narrative intervention and outcome measures. 50% will complete outcome measures only.
Masking Description: Assigned group is not masked. All roles will know which group (narrative or usual care) the patient has been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Intervention Group (Experimental): Patients in the narrative intervention group will participate in an interview and the resulting narrative will be uploaded to the electronic medical record. This group will also complete outcome measures (questionnaires) and exit interview.
  Interventions: Behavioral: Narrative Intervention
- Usual Care Group (No Intervention): Patients in the usual care group will complete outcome measures (questionnaires) and exit interview only.

INTERVENTIONS:
Behavioral: Narrative Intervention — Research staff conducts an open-ended, audio-recorded interview with the patient about their illness and how this illness has affected their psycho-social-spiritual well-being. The investigators will use the interview transcription to create a meta-narrative, which is then uploaded to the electronic medical record and the patient's primary nurse is notified that it is available to read.
  Arms: Narrative Intervention Group

SUMMARY:
Disparities in palliative care for patients with serious illness exist because of gaps in knowledge around patient centered psychological, social, and spiritual palliative care interventions. Patient-centered palliative care communication interventions must be informed by the perspectives of patients who are living each day with their serious illness. Yet, there is a lack of research about how to efficiently and effectively integrate the patient's narrative into the electronic health record (EHR). The central hypothesis of this proposal is that the implementation of a patient-centered narrative intervention with patients with serious illness will result in improved patient-nurse communication and improved patient psychosocial and spiritual well-being.

DETAILED DESCRIPTION:
The overall goal during this study will be to conduct a small scale pilot study with 80 hospitalized patients and 80 acute care nurses. Specific Aim 1 will establish acceptability, feasibility, and potential effect size of the patient-centered narrative intervention for hospitalized patients with serious illness. For specific aim 2, the investigators will compare the effects of the narrative intervention to usual care for the primary outcome of patient's perception of quality of communication and patient's psychosocial and spiritual well-being. For specific aim 3, the investigators will conduct usability testing, applying a user-task-system-environment evaluation process to determine essential requirements for integration and use of the patient-centered story into the EHR, from the perspective of an important end user: the acute-care bedside nurse. These results will support future R01 applications for testing/tailoring patient-centered narrative interventions to improve QoL for patients living with serious illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Has ability to read English.
* Capable of giving informed consent.
* Has diagnosis of at least one serious illness. For this study, the eligible diagnoses include: 1) New York Heart Class III or IV heart failure and/or 2) dialysis-dependent renal failure

Exclusion Criteria:

- None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Communication: QOC (Quality of Communication) survey | Time 1= Baseline, Time 2= 24-48 hours after baseline, Time 3- 24-48 hours after Time 2
  The QOC survey assesses patients' perceptions of the quality of communication with nurses. The QOC was initially developed from qualitative interviews and focus groups with diverse set of patients, families and providers. The QOC has 19 items, with scores ranging from 0 (worst) to 10 (best). Internal consistency reliability and construct validity of the QOC has been established across several illness groups, and the QOC survey's responsiveness to communication interventions has been demonstrated by changes in pre- and post-intervention scores.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)- 29 Profile | Time 1= Baseline, Time 2= 24-48 hours after baseline, Time 3- 24-48 hours after Time 2
  PROMIS- 29 profile v2.0 form (29 items), which assesses physiological, social, and psychological outcomes. These biopsychosocial domains include physical function, anxiety, depression, fatigue, sleep, ability to participate in social roles/activities, pain interference and intensity. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity. High scores represent more of the domain being measured. Thus, on symptom-oriented domains of PROMIS-29 (anxiety, depression, fatigue, pain interference, and sleep disturbance), higher scores represent worse symptomatology. On the function-oriented domains (physical functioning and social role) higher scores represent better functioning. For example, a high sleep disturbance score indicates high levels of sleep disturbance; a high physical functioning score indicates better physical function.
Change in Patient-Reported Outcome Measurement Information-System (PROMIS)- Psychosocial Illness Impact | Time 1= Baseline, Time 2= 24-48 hours after baseline, Time 3- 24-48 hours after Time 2
  The PROMIS positive item bank measure (8 items) assesses positive psychosocial outcomes of illness.The PROMIS negative item bank measure (8 items) assesses the direct negative psychosocial effect of illness, distinct from general emotional distress. The item bank instructs participants to think about how their illness has affected them. The item bank uses the time frames: before your illness" and "since your illness". For adults, each question has five response options ranging in value from two to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question, range 16-40. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Psychosocial Illness Impact-Positive, a T-score of 60 is one standard deviation (SD) better than average. By comparison, a Psychosocial Illness Impact-Positive T-score of 40 is one SD worse than average.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Coats, PhD, APRN-BC, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The final data set will include de-identified self-reported demographic and behavioral data from self-report, questionnaires, and interviews. The de-identified data and associated documentation will be made available to the community of scientists interested in palliative care as described in "access criteria." Additionally, aggregate, de-identified results will be submitted to ClinicalTrials.gov no later than one year after the trial's primary completion date.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to ten years
Access Criteria: The data and associated documentation will be made available to users only under a data-sharing agreement that provides for (a) a commitment to using the data only for research purposes and not to identify any individual patient; (b) a commitment to securing the data using appropriate computer technology; and (c) a commitment to destroying or returning the data after analyses are completed. Such a data-use agreement will be executed through the PI. The database of demographic and patient reported outcomes and de-identified transcripts will only be accessed via the investigator's secure website or shared via encrypted delivery.

REFERENCES:
- [Derived] Coats H, Shive N, Adrian B, Doorenbos AZ, Schmiege SJ. Integration of Person-Centered Narratives Into the Electronic Health Record. Nurs Res. 2023 Nov-Dec 01;72(6):421-429. doi: 10.1097/NNR.0000000000000680. Epub 2023 Aug 3. PMID 37582297
- [Derived] Coats H, Shive N, Doorenbos AZ, Schmiege SJ. Integration of Person-Centered Narratives Into the Electronic Health Record: Study Protocol. Nurs Res. 2020 Nov/Dec;69(6):483-489. doi: 10.1097/NNR.0000000000000463. PMID 32740306

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT04118569/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04118569/ICF_001.pdf